CLINICAL TRIAL: NCT06624930
Title: A Randomized Controlled Trial Adding Behavioural Counselling to Supervised Physical Activity in Cancer Survivors
Brief Title: Behaviour Change for Cancer Survivors Trial
Acronym: BOOST-Up
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Toronto Rehabilitation Institute (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Linda Trinh, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 518666
Record Dates: First submitted 2024-09-09; First posted 2024-10-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Exercise
Keywords: Cancer; Exercise
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: two group, parallel randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will be blinded to group assignment. Coordinating Research Assistants (RAs) will be the primary individuals responsible for scheduling all data collection assessments.
  The participants will attempt to book all 3 assessments with same RA assessor who meets the following criteria:
  * Are not a Qualified Exercise Professional (QEP) delivering one-on-one behavioural counselling
  * Are not a QEP that is running group webinar will not be involved in any data collection
  * Are not aware of participant's group allocation
  At the beginning of all data collection sessions, participants will be reminded not to disclose their any information about the activities performed for the study group assignment to the study assessor (RA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity + Behavioural Counselling (PA + BC) (Experimental): The PA+BC group will be given an individualized, home-based aerobic and resistance prescription based on baseline assessment and previous work. The participants will also receive behavioural counselling support sessions with a QEP every two weeks during the intervention period (12 total). The focus of these sessions will incorporate tailored behaviour change content from the M-PAC framework. At the end of the 6-month program, an individualized PA prescription will be provided based on their fitness level (adjusted throughout) to continue achieving the PA goal for the 6-month post intervention and 1-year post intervention follow-up.
  Interventions: Other: Behavioural Counselling
- Physical Activity + Exercise Couselling (PA + EC) (Active Comparator): The PA+EC group will be given an individualized, home-based aerobic and resistance prescription based on baseline assessment and previous work. The participants will also receive the same frequency of group-based and 1:1 counseling support sessions via Zoom as PA+BC participants. The focus of these sessions will be on exercise training principles for proper PA technique, how to monitor intensity, and progress PA safely to achieve the PA guidelines. The support sessions will be 30-45 minutes and delivered via Zoom each week in either group or 1:1 format depending on the topic.
  Interventions: Other: Exercise Counselling

INTERVENTIONS:
Other: Behavioural Counselling — The PA+BC group will receive a behavioural counselling support session with a QEP every two weeks during the intervention period (12 total). Of the 12 video-conferencing calls, one session will target reflective processes (instrumental/affective attitudes), five sessions will target behavioural regulation (action planning, coping planning, social support, goal setting), and four sessions will target reflexive processing (self-regulation, habit). The remaining two sessions are "booster sessions" to revisit topics discussed. The importance of sustaining PA for clinical outcomes (e.g., fatigue) and PA logs will be stressed. At the end of the 6-month program, an individualized PA prescription will be provided based on their fitness level (adjusted throughout) to continue achieving the PA goal for the 6-month post intervention and 1-year post intervention follow-up.
  Arms: Physical Activity + Behavioural Counselling (PA + BC)
Other: Exercise Counselling — The PA+EC group will receive the same frequency of group-based and 1:1 counseling support sessions via Zoom as PA+BC participants. However, the focus will be on exercise training principles for proper PA technique, how to monitor intensity, and progress PA safely to achieve the PA guidelines.
  Arms: Physical Activity + Exercise Couselling (PA + EC)

SUMMARY:
This study will be a two-arm RCT, to examine the effects of an entirely virtual, 6-month supervised PA program plus standard exercise counselling (PA+EC) versus a supervised PA plus motivationally-enhanced behavioral counselling (PA+BC) on moderate to vigorous physical activity (MVPA) in cancer survivors. A 6-month post intervention follow-up (T2) and 1-year post intervention follow-up (T3; 1-year follow-up from post-intervention) will take place after the intervention to address maintenance. The intervention is designed using evidence-based research in the fields of exercise oncology using effective clinical design and theoretical approaches, including behaviour change techniques, to gradually increase MVPA to at least 90 minutes per week in cancer survivors as per the exercise guidelines for cancer survivors.

DETAILED DESCRIPTION:
Many cancer survivors suffer from long-term side effects well beyond treatment such as fatigue, depression, muscle loss, which contributes to poor quality of life (QoL). Physical activity (PA) has a positive impact on clinical outcomes including improvements in overall QoL, cancer-specific mortality, and reducing treatment-related toxicities. Despite these benefits, the majority of cancer survivors, like their non-cancer counterparts, are not meeting public health PA guidelines. With COVID-19 restrictions easing, the health impact of the new normal may be long-lasting as cancer survivors have higher morbidity and mortality after contracting COVID-19. However, cancer survivors are realizing that they can receive quality and engaging access to care virtually in real-time to self-manage their symptoms. This represents a unique opportunity to test and deliver distance-based interventions in both clinical supportive cancer care and research trials. Short-term supervised PA programs can improve fitness and participant-reported outcomes in cancer survivors, but PA declines significantly post-treatment and long-term adherence is often low. This may also be due to the lack of available programming and facility-based, supervised programs that are easy to access even when they do exist. To achieve long-term health benefits, behaviour change must be sustained. Behaviour change interventions are complex with numerous interacting components that are often poorly described, especially with regard to how maintenance is defined. This hinders the understanding of intervention components that might facilitate PA maintenance. Behaviour change interventions improve PA over the course of the intervention; however, PA declines are more pronounced as the length of time between follow-up assessments increase. Nevertheless, the inclusion of theoretical components increases the likelihood of behaviour change in these interventions.

Recent PA guidelines for cancer survivors suggest 90 minutes of moderate-to-vigorous PA (MVPA) per week, and at least 2 days of strength training per week to accrue clinical benefits. PA-related benefits are only realized if cancer survivors adhere to and maintain PA. However, 74.8% and 86.1% of cancer survivors are not currently meeting aerobic PA and combined PA guidelines, respectively. Given that cancer survivors face several barriers to engaging in in-person PA (e.g., distance from clinical/community programs, treatment-related side effects ), there is a need to develop and assess the efficacy of distance-based approaches. The quality and effectiveness of distance-based interventions relative to non-telehealth home-based exercise or rehabilitation interventions are still unclear. Theoretical approaches to identifying key motivational outcomes to facilitate the adoption and maintenance of PA are limited. Behaviour change techniques such as self-monitoring, goal setting, social support, and action planning are shown to be effective techniques. Interventions that have used behavioural theory in cancer populations produced the largest overall effect size for behaviour change. However, little is known about which intervention mediators (e.g., behaviour change techniques) are responsible for long-term PA adherence.

The dominant theoretical approach in PA and cancer survivorship studies are social cognitive theories. While informative, theories rarely focus on maintenance through enacting on intention-behaviour gap mechanisms. The Multi-process Action Control (M-PAC) framework has a causal structure where an individual moves from intention formation to adoption of action control and onto maintenance of action control. According to the M-PAC, reflective processes (i.e., instrumental attitudes [expected benefits from performing PA], affective judgements [expected pleasure from performing PA], perceived capability [one's ability to perform PA] and perceived opportunity [perceived social/environmental circumstances to perform PA) are necessary for PA intention formation in cancer survivors. When these expectations are strong and positive, they culminate in the formation of PA intention (i.e., decision to enact regular PA). The dominant determinant when beginning regular PA is marked by the enactment of regulatory processes. Regulatory processes represent the behavioural, cognitive, and affective regulation strategies (e.g., planning, monitoring, attention focus) that are enacted to translate intention into PA. Finally, reflexive processes (i.e., habit [learned cue-behavior associations] and identity [role self-categorization] are those constructs that develop as a consequence of repeated successful behavioural outcomes over time. Therefore, while the M-PAC represents reflective, regulatory, and reflexive processes that build upon each other over time, each is expected to have some mediated feedback onto PA along with their own independent effect. Taken together, behaviour change is the product of reflective, regulatory, and reflexive processes that have facilitated an initial intention into successful on-going behaviour.

This proposal will address gaps in the PA maintenance literature to demonstrate: (1) changes in absolute values across behavioural performance of cancer survivors, (2) an increase in their magnitude of effect on PA over time; and (3) sex and gender differences in PA maintenance.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Confirmed diagnosis of cancer of any type (Stages I to III; localized)
* Have completed primary cancer treatment within 5 years
* At least 12 weeks after surgery completion
* At least 6 weeks after radiation treatment
* Proficient in English
* Physically inactive (self-report less than 90 min of MVPA/week )
* Ambulate in daily life with minimal gait aid use
* Access to a smartphone/tablet/computer with webcam for videoconferencing and a Bluetooth connection
* Access to the internet
* No cardiac contraindications (e.g., unstable angina, heart failure, coronary artery disease, diagnosed abnormality of heart rhythm)

Exclusion Criteria:

* A medical condition that prohibits PA (e.g., joint restriction or weight bearing precautions)
* Uncontrolled comorbidities or cardiovascular contraindications that would increase risk associated with supervised and unsupervised exercise (e.g., cardiac contraindications, severe arthritis, recent fall within the last 6-12 months)
* Presence of advanced cancer (i.e., Stage IV; metastatic)
* Pregnancy
* Do not intend to live in Canada for the next 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-Vigorous Physical Activity | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  Changes in MVPA will be assessed by accelerometry (ActiGraph Inc., Pensacola, FL.; model GT3X +). Participants will be mailed an accelerometer to wear on their right hip, fastened to a belt worn around the waist. The accelerometer will be worn during waking hours for 7 days, except when bathing or swimming.

SECONDARY OUTCOMES:
6-Minute Walk Test | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  6-minute walk test for aerobic endurance; from the Senior Fitness Test . Further distance walked indicates better physical function.
30-s Chair Stand Test | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  30-s chair stand test for lower body strength; from the Senior Fitness Test . Higher scores indicates better physical function.
Self-reported Physical Activity | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  Physical activity will be measured using a modified version of the (GLTEQ) Godin-Leisure Time Exercise Questionnaire 66 . This measure asks participants to self-report the frequency and duration of light, moderate, vigorous aerobic PA and resistance training for a typical week.
Functional Assessment of Cancer Therapy-General | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  Quality of life will be assessed by the validated Functional Assessment of Cancer Therapy-General (FACT-G) which consists of physical well-being (PWB), functional well-being (FWB), emotional well-being (EWB), and social well-being (SWB). 75
FACT-Fatigue | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  Fatigue will be assessed by the validated FACT-Fatigue (FACT-F) scale which includes the 27 items from the FACT-G scale plus the 13-item fatigue subscale.
Reflective, Regulatory, and Reflexive Processes | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  Standard measures from the M-PAC framework will be assessed including reflective processes of attitudes, and perceived capability and opportunity on a 7-point bipolar Likert scale.
Health Service Utilization Inventory | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  Health Economics Evaluation-Costs will be tracked using the Health Service Utilization Inventory with the view of conducting a cost-effectiveness analysis. The incremental cost of the intervention will be estimated and compared to changes in utility values converted from EQ5D results to evaluate the incremental cost per quality-adjusted life year of PA+BC. This study will be conducted from the perspective of the Canadian public healthcare payer and the participant. This inventory will be partially completed by each participant as well as members of the research team. Participants will complete the Health-Service Utilization Inventory and the research team will complete the iMTA Productivity Cost Questionnaire.
iMTA Productivity Cost Questionaire | T0 (Baseline), T1 (Mid-Point), T2 (Post-Intervention 6-Months), T3 (6-Month Follow Up After Intervention), T4 (1-Year Follow Up After Intervention)
  Health Economics Evaluation-Costs will be tracked using the iMTA Productivity Cost Questionnaire with the view of conducting a cost-effectiveness analysis. The incremental cost of the intervention will be estimated and compared to changes in utility values converted from EQ5D results to evaluate the incremental cost per quality-adjusted life year of PA+BC. This study will be conducted from the perspective of the Canadian public healthcare payer and the participant. This inventory will be partially completed by each participant as well as members of the research team. Participants will complete the Health-Service Utilization Inventory and the research team will complete the iMTA Productivity Cost Questionnaire.
Age | Baseline (T0)
  Demographic variable of age will be assessed. Units of measurement is years.
Sex | Baseline (T0)
  Demographic variable of biological sex will be assessed. Response options are; male and female.
Gender | Baseline (T0)
  Demographic variable of gender will be assessed. Response options include; male, female, and other (self-reported).
Marital status | Baseline (T0)
  Demographic variable of marital status will be assessed. Response options are; single, married, common-law, separated, widowed, and divorced.
Highest Level of Education | Baseline (T0)
  Demographic variable of highest level of education will be assessed. Response options are; some high school, completed high school, some university/college, completed university/college, some graduate school, completed graduate school.
Current Employment Status | Baseline (T0)
  Demographic variable of current employment status will be assessed. Response options are; disability, retired, part-time, homemaker, full-time, and unemployed.
Ethnicity | Baseline (T0)
  Demographic variable of ethnicity will be assessed. Response options are; White, Chinese, South Asian, Black, Filipino, Latin American, South East Asian, Arab, West Asian, Korean, Japanese, and other.
Body Mass Index | Baseline (T0)
  Demographic variable of body mass index will be assessed. Units of measurement are height (ft.) and weight (lb.). Weight and height will be combined to report BMI in kg/m^2.
Medical Demographics | Baseline (T0)
  Medical variables include: cancer type, date of diagnosis, cancer stage, cancer spread, treatment, current status, recurrences, presence of side effects, impact of cancer on physical activity, comorbidities and current disease status.
Gender Index | Baseline (T0)
  The Gender Index will be used to assess gender associated risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Trinh, PhD, Principal Investigator — University of Toronto
Locations (1):
- Exercise Oncology Lab - University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Cancer Statistics Advisory Committee in collaboration with the Canadian Cancer Society SC and the PHA of C. Canadian Cancer Statistics 2021.; 2021.
- [Background] Patel AV, Friedenreich CM, Moore SC, Hayes SC, Silver JK, Campbell KL, Winters-Stone K, Gerber LH, George SM, Fulton JE, Denlinger C, Morris GS, Hue T, Schmitz KH, Matthews CE. American College of Sports Medicine Roundtable Report on Physical Activity, Sedentary Behavior, and Cancer Prevention and Control. Med Sci Sports Exerc. 2019 Nov;51(11):2391-2402. doi: 10.1249/MSS.0000000000002117. PMID 31626056
- [Background] Gerritsen JK, Vincent AJ. Exercise improves quality of life in patients with cancer: a systematic review and meta-analysis of randomised controlled trials. Br J Sports Med. 2016 Jul;50(13):796-803. doi: 10.1136/bjsports-2015-094787. Epub 2015 Dec 30. PMID 26719503
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Mishra SI, Scherer RW, Snyder C, Geigle PM, Berlanstein DR, Topaloglu O. Exercise interventions on health-related quality of life for people with cancer during active treatment. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD008465. doi: 10.1002/14651858.CD008465.pub2. PMID 22895974
- [Background] Patel AV, Bernstein L, Deka A, Feigelson HS, Campbell PT, Gapstur SM, Colditz GA, Thun MJ. Leisure time spent sitting in relation to total mortality in a prospective cohort of US adults. Am J Epidemiol. 2010 Aug 15;172(4):419-29. doi: 10.1093/aje/kwq155. Epub 2010 Jul 22. PMID 20650954
- [Background] Thraen-Borowski KM, Gennuso KP, Cadmus-Bertram L. Accelerometer-derived physical activity and sedentary time by cancer type in the United States. PLoS One. 2017 Aug 14;12(8):e0182554. doi: 10.1371/journal.pone.0182554. eCollection 2017. PMID 28806753
- [Background] Tabaczynski A, Bastas D, Whitehorn A, Trinh L. Changes in physical activity and associations with quality of life among a global sample of cancer survivors during the COVID-19 pandemic. J Cancer Surviv. 2023 Aug;17(4):1191-1201. doi: 10.1007/s11764-021-01156-x. Epub 2022 Jan 26. PMID 35079964
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Lopez CJ, Edwards B, Langelier DM, Chang EK, Chafranskaia A, Jones JM. Delivering Virtual Cancer Rehabilitation Programming During the First 90 Days of the COVID-19 Pandemic: A Multimethod Study. Arch Phys Med Rehabil. 2021 Jul;102(7):1283-1293. doi: 10.1016/j.apmr.2021.02.002. Epub 2021 Feb 19. PMID 33617864
- [Background] Courneya KS, Segal RJ, Gelmon K, Reid RD, Mackey JR, Friedenreich CM, Proulx C, Lane K, Ladha AB, Vallance JK, McKenzie DC. Predictors of supervised exercise adherence during breast cancer chemotherapy. Med Sci Sports Exerc. 2008 Jun;40(6):1180-7. doi: 10.1249/MSS.0b013e318168da45. PMID 18460985
- [Background] Bluethmann SM, Vernon SW, Gabriel KP, Murphy CC, Bartholomew LK. Taking the next step: a systematic review and meta-analysis of physical activity and behavior change interventions in recent post-treatment breast cancer survivors. Breast Cancer Res Treat. 2015 Jan;149(2):331-42. doi: 10.1007/s10549-014-3255-5. Epub 2015 Jan 3. PMID 25555831
- [Background] Blaney JM, Lowe-Strong A, Rankin-Watt J, Campbell A, Gracey JH. Cancer survivors' exercise barriers, facilitators and preferences in the context of fatigue, quality of life and physical activity participation: a questionnaire-survey. Psychooncology. 2013 Jan;22(1):186-94. doi: 10.1002/pon.2072. Epub 2011 Oct 6. PMID 23296635
- [Background] Grimmett C, Corbett T, Brunet J, Shepherd J, Pinto BM, May CR, Foster C. Systematic review and meta-analysis of maintenance of physical activity behaviour change in cancer survivors. Int J Behav Nutr Phys Act. 2019 Apr 27;16(1):37. doi: 10.1186/s12966-019-0787-4. PMID 31029140
- [Background] Rhodes RE, Sui W. Physical Activity Maintenance: A Critical Narrative Review and Directions for Future Research. Front Psychol. 2021 Sep 6;12:725671. doi: 10.3389/fpsyg.2021.725671. eCollection 2021. PMID 34552537
- [Background] McEwan D, Rhodes RE, Beauchamp MR. What Happens When the Party is Over?: Sustaining Physical Activity Behaviors after Intervention Cessation. Behav Med. 2022 Jan-Mar;48(1):1-9. doi: 10.1080/08964289.2020.1750335. Epub 2020 Apr 10. PMID 32275199
- [Background] Rhodes RE. Multi-Process Action Control in Physical Activity: A Primer. Front Psychol. 2021 Dec 15;12:797484. doi: 10.3389/fpsyg.2021.797484. eCollection 2021. PMID 34975698
- [Background] Kessels E, Husson O, van der Feltz-Cornelis CM. The effect of exercise on cancer-related fatigue in cancer survivors: a systematic review and meta-analysis. Neuropsychiatr Dis Treat. 2018 Feb 9;14:479-494. doi: 10.2147/NDT.S150464. eCollection 2018. PMID 29445285
- [Background] Groen WG, van Harten WH, Vallance JK. Systematic review and meta-analysis of distance-based physical activity interventions for cancer survivors (2013-2018): We still haven't found what we're looking for. Cancer Treat Rev. 2018 Sep;69:188-203. doi: 10.1016/j.ctrv.2018.07.012. Epub 2018 Jul 21. PMID 30077954
- [Background] Schmitz KH, Campbell AM, Stuiver MM, Pinto BM, Schwartz AL, Morris GS, Ligibel JA, Cheville A, Galvao DA, Alfano CM, Patel AV, Hue T, Gerber LH, Sallis R, Gusani NJ, Stout NL, Chan L, Flowers F, Doyle C, Helmrich S, Bain W, Sokolof J, Winters-Stone KM, Campbell KL, Matthews CE. Exercise is medicine in oncology: Engaging clinicians to help patients move through cancer. CA Cancer J Clin. 2019 Nov;69(6):468-484. doi: 10.3322/caac.21579. Epub 2019 Oct 16. PMID 31617590
- [Background] Ibeggazene S, Turner R, Rosario D, Bourke L. Remote interventions to improve exercise behaviour in sedentary people living with and beyond cancer: a systematic review and meta-analysis. BMC Cancer. 2021 Mar 24;21(1):308. doi: 10.1186/s12885-021-07989-0. PMID 33761906
- [Background] Goode AD, Lawler SP, Brakenridge CL, Reeves MM, Eakin EG. Telephone, print, and Web-based interventions for physical activity, diet, and weight control among cancer survivors: a systematic review. J Cancer Surviv. 2015 Dec;9(4):660-82. doi: 10.1007/s11764-015-0442-2. Epub 2015 Mar 11. PMID 25757733
- [Background] Roberts AL, Fisher A, Smith L, Heinrich M, Potts HWW. Digital health behaviour change interventions targeting physical activity and diet in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2017 Dec;11(6):704-719. doi: 10.1007/s11764-017-0632-1. Epub 2017 Aug 4. PMID 28779220
- [Background] Finlay A, Wittert G, Short CE. A systematic review of physical activity-based behaviour change interventions reaching men with prostate cancer. J Cancer Surviv. 2018 Aug;12(4):571-591. doi: 10.1007/s11764-018-0694-8. Epub 2018 May 16. PMID 29770953
- [Background] Stacey FG, James EL, Chapman K, Courneya KS, Lubans DR. A systematic review and meta-analysis of social cognitive theory-based physical activity and/or nutrition behavior change interventions for cancer survivors. J Cancer Surviv. 2015 Jun;9(2):305-38. doi: 10.1007/s11764-014-0413-z. Epub 2014 Nov 29. PMID 25432633
- [Background] Pudkasam S, Polman R, Pitcher M, Fisher M, Chinlumprasert N, Stojanovska L, Apostolopoulos V. Physical activity and breast cancer survivors: Importance of adherence, motivational interviewing and psychological health. Maturitas. 2018 Oct;116:66-72. doi: 10.1016/j.maturitas.2018.07.010. Epub 2018 Jul 23. PMID 30244781
- [Background] Paterson C, Bacon R, Dwyer R, Morrison KS, Toohey K, O'Dea A, Slade J, Mortazavi R, Roberts C, Pranavan G, Cooney C, Nahon I, Hayes SC. The Role of Telehealth During the COVID-19 Pandemic Across the Interdisciplinary Cancer Team: Implications for Practice. Semin Oncol Nurs. 2020 Dec;36(6):151090. doi: 10.1016/j.soncn.2020.151090. Epub 2020 Oct 15. PMID 33218886
- [Background] Hailey V, Rojas-Garcia A, Kassianos AP. A systematic review of behaviour change techniques used in interventions to increase physical activity among breast cancer survivors. Breast Cancer. 2022 Mar;29(2):193-208. doi: 10.1007/s12282-021-01323-z. Epub 2022 Jan 6. PMID 34989962
- [Background] Faro JM, Mattocks KM, Nagawa CS, Lemon SC, Wang B, Cutrona SL, Sadasivam RS. Physical Activity, Mental Health, and Technology Preferences to Support Cancer Survivors During the COVID-19 Pandemic: Cross-sectional Study. JMIR Cancer. 2021 Feb 3;7(1):e25317. doi: 10.2196/25317. PMID 33471776
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Feasibility and preliminary efficacy of adding behavioral counseling to supervised physical activity in kidney cancer survivors: a randomized controlled trial. Cancer Nurs. 2014 Sep-Oct;37(5):E8-22. doi: 10.1097/NCC.0b013e3182a40fb6. PMID 24232192
- [Background] Trinh L, Kramer AF, Rowland K, Strom DA, Wong JN, McAuley E. A pilot feasibility randomized controlled trial adding behavioral counseling to supervised physical activity in prostate cancer survivors: behavior change in prostate cancer survivors trial (BOOST). J Behav Med. 2021 Apr;44(2):172-186. doi: 10.1007/s10865-020-00185-8. Epub 2020 Sep 26. PMID 32979134
- [Background] Marcus BH, Dubbert PM, Forsyth LH, McKenzie TL, Stone EJ, Dunn AL, Blair SN. Physical activity behavior change: issues in adoption and maintenance. Health Psychol. 2000 Jan;19(1S):32-41. doi: 10.1037/0278-6133.19.suppl1.32. PMID 10709946
- [Background] Rogers LQ, Courneya KS, Anton PM, Hopkins-Price P, Verhulst S, Vicari SK, Robbs RS, Mocharnuk R, McAuley E. Effects of the BEAT Cancer physical activity behavior change intervention on physical activity, aerobic fitness, and quality of life in breast cancer survivors: a multicenter randomized controlled trial. Breast Cancer Res Treat. 2015 Jan;149(1):109-19. doi: 10.1007/s10549-014-3216-z. Epub 2014 Nov 23. PMID 25417174
- [Background] Oberoi S, Robinson PD, Cataudella D, Culos-Reed SN, Davis H, Duong N, Gibson F, Gotte M, Hinds P, Nijhof SL, Tomlinson D, van der Torre P, Cabral S, Dupuis LL, Sung L. Physical activity reduces fatigue in patients with cancer and hematopoietic stem cell transplant recipients: A systematic review and meta-analysis of randomized trials. Crit Rev Oncol Hematol. 2018 Feb;122:52-59. doi: 10.1016/j.critrevonc.2017.12.011. Epub 2017 Dec 16. PMID 29458789
- [Background] Bluethmann SM, Bartholomew LK, Murphy CC, Vernon SW. Use of Theory in Behavior Change Interventions. Health Educ Behav. 2017 Apr;44(2):245-253. doi: 10.1177/1090198116647712. Epub 2016 Jul 10. PMID 27226430
- [Background] Kwasnicka D, Dombrowski SU, White M, Sniehotta F. Theoretical explanations for maintenance of behaviour change: a systematic review of behaviour theories. Health Psychol Rev. 2016 Sep;10(3):277-96. doi: 10.1080/17437199.2016.1151372. Epub 2016 Mar 7. PMID 26854092
- [Background] Rhodes RE, de Bruijn GJ. How big is the physical activity intention-behaviour gap? A meta-analysis using the action control framework. Br J Health Psychol. 2013 May;18(2):296-309. doi: 10.1111/bjhp.12032. PMID 23480428
- [Background] Rhodes RE, Yao CA. Models accounting for intention-behavior discordance in the physical activity domain: a user's guide, content overview, and review of current evidence. Int J Behav Nutr Phys Act. 2015 Feb 7;12:9. doi: 10.1186/s12966-015-0168-6. PMID 25890238
- [Background] Vallerand JR, Rhodes RE, Walker GJ, Courneya KS. Feasibility and preliminary efficacy of an exercise telephone counseling intervention for hematologic cancer survivors: a phase II randomized controlled trial. J Cancer Surviv. 2018 Jun;12(3):357-370. doi: 10.1007/s11764-018-0675-y. Epub 2018 Feb 6. PMID 29411314
- [Background] Tabaczynski A, Arbour-Nicitopoulos KP, Rhodes RE, Sabiston CM, Trinh L. Correlates of Physical Activity Participation among Individuals Diagnosed with Cancer: An Application of the Multi-Process Action Control Framework. Int J Environ Res Public Health. 2023 Feb 28;20(5):4345. doi: 10.3390/ijerph20054345. PMID 36901355
- [Background] Volz SC, Furman CR, Rothman AJ. Psychological Correlates of Perceived Physical Activity Engagement During the COVID-19 Pandemic Among Previously Active Individuals. Behav Med. 2023 Jan-Mar;49(1):7-14. doi: 10.1080/08964289.2021.1929811. Epub 2021 Oct 26. PMID 34702131
- [Background] Rhodes RE, Liu S, Lithopoulos A, Zhang CQ, Garcia-Barrera MA. Correlates of Perceived Physical Activity Transitions during the COVID-19 Pandemic among Canadian Adults. Appl Psychol Health Well Being. 2020 Dec;12(4):1157-1182. doi: 10.1111/aphw.12236. Epub 2020 Oct 1. PMID 33006279
- [Background] Elshahat S, Treanor C, Donnelly M. Factors influencing physical activity participation among people living with or beyond cancer: a systematic scoping review. Int J Behav Nutr Phys Act. 2021 Apr 6;18(1):50. doi: 10.1186/s12966-021-01116-9. PMID 33823832
- [Background] Coughlin SS, Stewart J. Use of Consumer Wearable Devices to Promote Physical Activity: A Review of Health Intervention Studies. J Environ Health Sci. 2016 Nov;2(6):10.15436/2378-6841.16.1123. doi: 10.15436/2378-6841.16.1123. Epub 2016 Nov 30. PMID 28428979
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Wright CE, Rhodes RE, Ruggiero EW, Sheeran P. Benchmarking the effectiveness of interventions to promote physical activity: A metasynthesis. Health Psychol. 2021 Nov;40(11):811-821. doi: 10.1037/hea0001118. PMID 34914485
- [Background] Ormel HL, van der Schoot GGF, Sluiter WJ, Jalving M, Gietema JA, Walenkamp AME. Predictors of adherence to exercise interventions during and after cancer treatment: A systematic review. Psychooncology. 2018 Mar;27(3):713-724. doi: 10.1002/pon.4612. Epub 2018 Jan 26. PMID 29247584
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Vallerand JR, Rhodes RE, Walker GJ, Courneya KS. Correlates of meeting the combined and independent aerobic and strength exercise guidelines in hematologic cancer survivors. Int J Behav Nutr Phys Act. 2017 Mar 28;14(1):44. doi: 10.1186/s12966-017-0498-7. PMID 28351397
- [Background] Rhodes RE, Lithopoulos A. The Physical Activity Regulation Scale: Development and validity testing. Health Psychol. 2023 Jun;42(6):378-387. doi: 10.1037/hea0001283. PMID 37227880
- [Background] Gardner B, Abraham C, Lally P, de Bruijn GJ. Towards parsimony in habit measurement: testing the convergent and predictive validity of an automaticity subscale of the Self-Report Habit Index. Int J Behav Nutr Phys Act. 2012 Aug 30;9:102. doi: 10.1186/1479-5868-9-102. PMID 22935297
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Correlates of physical activity in a population-based sample of kidney cancer survivors: an application of the theory of planned behavior. Int J Behav Nutr Phys Act. 2012 Aug 6;9:96. doi: 10.1186/1479-5868-9-96. PMID 22866956
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J. The Functional Assessment of Cancer Therapy Scale: Development and Validation of the General Measure. J Clin Oncol. 2023 Dec 10;41(35):5335-5344. doi: 10.1200/JCO.22.02775. PMID 38056080
- [Background] Brucker PS, Yost K, Cashy J, Webster K, Cella D. General population and cancer patient norms for the Functional Assessment of Cancer Therapy-General (FACT-G). Eval Health Prof. 2005 Jun;28(2):192-211. doi: 10.1177/0163278705275341. PMID 15851773
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Day S, Mason R, Tannenbaum C, Rochon PA. Essential metrics for assessing sex & gender integration in health research proposals involving human participants. PLoS One. 2017 Aug 30;12(8):e0182812. doi: 10.1371/journal.pone.0182812. eCollection 2017. PMID 28854192
- [Background] Pelletier R, Ditto B, Pilote L. A composite measure of gender and its association with risk factors in patients with premature acute coronary syndrome. Psychosom Med. 2015 Jun;77(5):517-26. doi: 10.1097/PSY.0000000000000186. PMID 25984818
- [Background] Pilote L, Karp I. GENESIS-PRAXY (GENdEr and Sex determInantS of cardiovascular disease: From bench to beyond-Premature Acute Coronary SYndrome). Am Heart J. 2012 May;163(5):741-746.e2. doi: 10.1016/j.ahj.2012.01.022. PMID 22607849
- [Background] Norris CM, Johnson NL, Hardwicke-Brown E, McEwan M, Pelletier R, Pilote L. The Contribution of Gender to Apparent Sex Differences in Health Status Among Patients with Coronary Artery Disease. J Womens Health (Larchmt). 2017 Jan;26(1):50-57. doi: 10.1089/jwh.2016.5744. Epub 2016 Jul 11. PMID 27400270
- [Background] Rhodes RE, Beauchamp MR, Quinlan A, Symons Downs D, Warburton DER, Blanchard CM. Predicting the physical activity of new parents who participated in a physical activity intervention. Soc Sci Med. 2021 Sep;284:114221. doi: 10.1016/j.socscimed.2021.114221. Epub 2021 Jul 10. PMID 34274708
- [Background] Bouwmans C, Krol M, Severens H, Koopmanschap M, Brouwer W, Hakkaart-van Roijen L. The iMTA Productivity Cost Questionnaire: A Standardized Instrument for Measuring and Valuing Health-Related Productivity Losses. Value Health. 2015 Sep;18(6):753-8. doi: 10.1016/j.jval.2015.05.009. Epub 2015 Aug 20. PMID 26409601
- [Background] Xie F, Pullenayegum E, Gaebel K, Bansback N, Bryan S, Ohinmaa A, Poissant L, Johnson JA; Canadian EQ-5D-5L Valuation Study Group. A Time Trade-off-derived Value Set of the EQ-5D-5L for Canada. Med Care. 2016 Jan;54(1):98-105. doi: 10.1097/MLR.0000000000000447. PMID 26492214
- [Derived] Trinh L, Rhodes RE, Alibhai SMH, Campbell KL, Langelier DM, Chang E, Colella T, Chan B, Santa Mina D, Oh P, McAuley E. A randomized controlled trial adding behavioral counseling to supervised physical activity in people living with and beyond cancer (BOOST-UP-): a study protocol for a live remotely-delivered behavior change intervention. BMC Cancer. 2025 May 9;25(1):847. doi: 10.1186/s12885-025-13904-8. PMID 40346460